CLINICAL TRIAL: NCT05781685
Title: The Influence of Testosterone on Experimental Pain Perception and Social Psychological Functioning
Brief Title: The Influence of Testosterone on Experimental Pain Perception
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: American Psychological Association (APA) (Other)
Responsible Party: Principal Investigator, Chance Strenth, Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1100595-3
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Acute Pain
Keywords: testosterone; pain tolerance; estradiol; progesterone
MeSH Terms: conditions — Acute Pain | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigational drug pharmacy providing the sublingual testosterone masked the drugs. Neither the participants nor the investigators knew who was receiving testosterone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Experimental): Sublingual testosterone
  Interventions: Drug: Testosterone; Other: Placebo Syrup
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Testosterone; Other: Placebo Syrup

INTERVENTIONS:
Drug: Testosterone — Sublingual testosterone was administered to participants. Participants would self-administer the testosterone to themselves.
Other: Placebo Syrup — Oil-based sublingual product.

SUMMARY:
This trial examined how the administration of exogenous testosterone would influence pain tolerance and other endogenous steroids (i.e. estradiol and progesterone).

ELIGIBILITY:
Inclusion Criteria:

* Healthy college-aged females that are over the age of 18 and younger than 25 will be used for this study.

Exclusion Criteria:

* The following criteria will exclude a participant from the study:
* Anyone that has a tree nut allergy.
* Women that are pregnant or may feel that they may be pregnant or breast-feeding.
* Anyone taking supplements that may influence their testosterone level.
* Anyone taking any kind of steroid that may increase their testosterone level.
* Anyone that smokes tobacco or uses smokeless tobacco.
* Anyone that reports any condition associated with nerve damage.
* Anyone that is using hormonal contraceptive.
* Anyone who was sick or unwell at the time of screening.
* Each participant completed a Testosterone Pre-Screen form. This form asked each participant individually whether they are taking any drugs or have any conditions that might be exacerbated by testosterone. This form was completed before they signed the consent form and each time they arrived in the lab for an experimental session.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone, Placebo: Sublingual testosterone
  First: Testosterone: Sublingual testosterone was administered to participants. Participants would self-administer the testosterone to themselves.
  Second: Placebo Syrup: Oil-based sublingual product.
- Placebo, Testosterone: Placebo
  First: Placebo Syrup: Oil-based sublingual product.
  Second: Testosterone: Sublingual testosterone was administered to participants. Participants would self-administer the testosterone to themselves.
Period: First Period of Intervention (Day 1)
Arm/Group | Testosterone, Placebo | Placebo, Testosterone
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Period of Intervention (Day 4)
Arm/Group | Testosterone, Placebo | Placebo, Testosterone
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone, Placebo | Placebo, Testosterone | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.8 (.92) | 18.6 (.97) | 18.7 (.92338)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Tolerance
Description: The ischemic discomfort task applied a sphygmomanometer (blood pressure cuff) 5 cm below their elbow. The cuff was inflated to 200 mmHg. Pain tolerance was measured by how long they could tolerate the ischemic discomfort task. However, task was only allowed to last for 6 minutes
Time Frame: 4 hours After Administration
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 20 | 20
Seconds | 224.20500 (91.144110) | 224.92615 (94.080395)

2. Secondary Outcome: Changes Testosterone Levels
Description: The measured testosterone levels in the participants before and after receiving the intervention
Time Frame: Prior to Intervention (Baseline), 15 minutes Post Intervention
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Placebo: Placebo
  Placebo Syrup: Oil-based sublingual product.
  Second: Testosterone: Sublingual testosterone was administered to participants. Participants would self-administer the testosterone to themselves.
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 20 | 20
pg/ml | 580.299600 (45.919951749402) | 38.3972 (10.859257363884)

3. Secondary Outcome: Changes Estradiol Levels
Description: The measured estradiol levels in the participants before and after receiving the intervention.
Time Frame: Prior to Intervention (Baseline), 15 minutes Post Intervention
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 20 | 20
pg/ml | -0.903160000000 (0.1943390807362) | 0.1801549999999 (0.0950549798844)

4. Secondary Outcome: Changes Progesterone Levels
Description: he measured progesterone levels in the participants before and after receiving the intervention.
Time Frame: Prior to Intervention (Baseline), 15 minutes Post Intervention
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 20 | 20
pg/ml | -423.63719 (72.274306309941) | 29.381135 (59.866738560717)

ADVERSE EVENTS:
Time Frame: From baseline approximately up to 3 months.
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT05781685/Prot_SAP_000.pdf